CLINICAL TRIAL: NCT03040960
Title: Risk Factors for Staphylococcus Aureus Surgical Site Infections in Orthopedic and Trauma Surgery
Acronym: ISO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC16.223; 1985246 (Other: CNIL)
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Staphylococcus Aureus; Surgical Wound Infection; Orthopedic Disorder; Traumatology
Keywords: infection; wound infection; surgical wound infection; Staphylococcal infections; wound and injuries; postoperative complications; Gram-positive bacterial infections; bacterial infections
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection; Musculoskeletal Diseases; Infections; Wound Infection; Wounds and Injuries; Postoperative Complications; Gram-Positive Bacterial Infections; Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The most commonly identified organism for Surgical Site Infection (SSI) in orthopedic surgery is Staphylococcus aureus but risk factors for mono microbial S.aureus SSI are not well-known. The aim of this study was to evaluated the incidence rate of S. aureus SSI over the years and risk factors of these infections in a french University Hospital.

DETAILED DESCRIPTION:
Surgical site infections (SSI) in orthopedic surgery are responsible for reduced quality of life, increased length of hospital stay and costs. The most commonly identified organism is Staphylococcus aureus but risk factors for mono microbial S.aureus SSI are not well-known.The aim of this study was to evaluate the incidence rate trend of S. aureus SSI over the years and risk factors of theses infections in a french University Hospital.

The knowledge obtained by this study will enable identification of the surgical patients most at risk of developping S. aureus SSI, and who would probably benefit most from new interventions given prophylactically and specifically to prevent S. aureus infections.

ELIGIBILITY:
Inclusion Criteria:

* orthopedic or traumatology surgeries performed in Grenoble University Hospital,
* from january 1st 2012 to april 30th 2015,
* the subject is undergoing one of the following surgical procedures : knee and hip arthroplasties, osteosynthesis of proximal femur and other osteosynthesis except skull and spine.
* the subject is 16 years of age or older

Exclusion Criteria:

* non orthopedic or trauma surgery performed in Grenoble University Hospital,
* spine surgeries,
* surgeries of the hand, scaphoid and carpal bones.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing orthopedic or traumatologiy surgeries in Grenoble university hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Risk factors of S. aureus surgical site infections. | up to 1 year following surgery
  univariate analysis of potential risk factors. Data with p value less than 0.1 were included in a logistic regression model

SECONDARY OUTCOMES:
The incidence rate trend of S. aureus SSI over the year. | from january 1st 2012 to april 30th 2015
  linear regression slope test of S. aureus SSI incidence rates by years

CONTACTS AND LOCATIONS:
Overall Officials: Caroline landelle, PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalmeijer MD, van Nieuwland-Bollen E, Bogaers-Hofman D, de Baere GA. Nasal carriage of Staphylococcus aureus is a major risk factor for surgical-site infections in orthopedic surgery. Infect Control Hosp Epidemiol. 2000 May;21(5):319-23. doi: 10.1086/501763. PMID 10823564
- [Background] Korol E, Johnston K, Waser N, Sifakis F, Jafri HS, Lo M, Kyaw MH. A systematic review of risk factors associated with surgical site infections among surgical patients. PLoS One. 2013 Dec 18;8(12):e83743. doi: 10.1371/journal.pone.0083743. eCollection 2013. PMID 24367612
- [Background] Marimuthu K, Eisenring MC, Harbarth S, Troillet N. Epidemiology of Staphylococcus aureus Surgical Site Infections. Surg Infect (Larchmt). 2016 Apr;17(2):229-35. doi: 10.1089/sur.2015.055. Epub 2015 Dec 31. PMID 26720215
- [Background] Lepelletier D, Saliou P, Lefebvre A, Lucet JC, Grandbastien B, Bruyere F, Stahl JP, Keita-Perse O, Berthelot P, Aho S; workgroup SF2H. "Preoperative risk management: strategy for Staphylococcus aureus preoperative decolonization" (2013 update). French society of Hospital Hygiene. Med Mal Infect. 2014 Jun;44(6):261-7. doi: 10.1016/j.medmal.2014.04.003. Epub 2014 May 14. No abstract available. PMID 24835378
- [Background] Webster J, Osborne S. Preoperative bathing or showering with skin antiseptics to prevent surgical site infection. Cochrane Database Syst Rev. 2015 Feb 20;2015(2):CD004985. doi: 10.1002/14651858.CD004985.pub5. PMID 25927093